CLINICAL TRIAL: NCT00069381
Title: Skills Training, Exposure, and Their Combination in Childhood Abuse PTSD
Brief Title: Treatment for Women With Post-Traumatic Stress Disorder Related to Childhood Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH062347 (NIH); R01MH062347 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2003-09-24; First posted 2003-09-25 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- study arm (Experimental)
  Interventions: Behavioral: Psychotherapy treatment

INTERVENTIONS:
Behavioral: Psychotherapy treatment

SUMMARY:
This study will compare one- and two-component treatments in women with post-traumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
PTSD is a debilitating and often chronic anxiety disorder with serious psychiatric comorbidity. The most common trauma associated with PTSD among women is childhood abuse. PTSD related to childhood abuse may cause problems with emotion regulation and interpersonal functioning. This study will address three domains of PTSD related to childhood abuse: emotion management problems, interpersonal problems, and PTSD symptoms.

Participants in this study will be randomly assigned to 16 sessions of one of three treatments: Skills Training for Affective and Interpersonal Regulation (STAIR), which focuses on helping individuals strengthen and build skills in managing feelings and improving interpersonal relationships; Modified Prolonged Exposure (MPE), which focuses on developing narratives of abuse history and completing an "emotional processing" of the trauma in a safe environment; and a combination of STAIR and MPE. Dropout rates and adverse effects will be measured.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for Post-Traumatic Stress Disorder related to childhood physical and/or sexual abuse by a care-giver
* At least one clear memory of the abuse
* Willing to have all assessments tape recorded and sessions video taped
* Willing to maintain any concurrent treatments for the duration of the study

Exclusion Criteria:

* Bipolar Disorder
* Eating Disorder
* Borderline Personality Disorder
* Active substance abuse or dependence
* Living with the abuser
* Self mutilation
* Pregnancy

Ages: 22 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2002-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
outcome | within study timeframe

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Child Study Center Institute for Trauma and Stress, New York, New York, United States

REFERENCES:
- [Derived] Cloitre M, Stovall-McClough KC, Nooner K, Zorbas P, Cherry S, Jackson CL, Gan W, Petkova E. Treatment for PTSD related to childhood abuse: a randomized controlled trial. Am J Psychiatry. 2010 Aug;167(8):915-24. doi: 10.1176/appi.ajp.2010.09081247. Epub 2010 Jul 1. PMID 20595411
- See also: Related Info — http://www.AboutOurKids.org